CLINICAL TRIAL: NCT00094380
Title: Treatment of Systemic Lupus Erythematosus With CTLA4-IgG4m Plus Cyclophosphamide: A Phase I/IIA Study
Brief Title: Treating Systemic Lupus Erythematosus (SLE) Patients With CTLA4-IgG4m (RG2077)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN002AI
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Nephritis
Keywords: SLE; Lupus; Systemic Lupus Erythematosus; Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclophosphamide

ARMS (3):
- Dose-escalation portion: Low dose CTLA4-IgG4m (RG2077) (Experimental): Three patients will receive a single intravenous infusion of 0.2 mg/kg CTLA4-IgG4m following the scheduled cyclophosphamide infusion on the same day. If one or more dose-limiting toxicities (CTC grade 3 or higher adverse event in the first 28 days after CTLA4-IgG4m administration that is possibly, probably, or definitely related to CTLA4-IgG4m (RG2077)). are observed, enrollment in the trial will be suspended pending DSMB review. If no dose-limiting toxicity is observed in the 0.2mg/kg dose, three patients will receive a single intravenous infusion of 2 mg/kg of CTLA4-IgG4m following the scheduled cyclophosphamide infusion on the same day. If one or more dose-limiting toxicities are observed, enrollment will be suspended pending review by the Data Safety and Monitoring Board (DSMB).If no dose-limiting toxicity is observed in the 2 mg/kg dose, treatment of patients with 10 mg/kg of CTLA4-IgG4m in combination with cyclophosphamide will proceed.
  Interventions: Drug: CTLA4-IgG4m (RG2077); Drug: Cyclophosphamide
- Part IIA: CTLA4-IgG4m (Experimental): Participants randomized to the CTLA4-IgG4m Arm will receive a single intravenous infusion of 10 mg/kg CTLA4-IgG4m (RG2077) following the scheduled cyclophosphamide infusion on the same day
  Interventions: Drug: CTLA4-IgG4m (RG2077); Drug: Cyclophosphamide
- Part IIA: Control Group (Experimental): Participants randomized to the control group will not receive treatment with CTLA4-IgG4m (RG2077); these participants will undergo all study evaluations with the exception of the CTLA4-IgG4m (RG2077) pharmacokinetic evaluations and immunogenicity evaluations.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CTLA4-IgG4m (RG2077)
  Arms: Dose-escalation portion: Low dose CTLA4-IgG4m (RG2077); Part IIA: CTLA4-IgG4m
Drug: Cyclophosphamide

SUMMARY:
The purpose of this study is to examine the safety of a single dose of RG2077 in patients with systemic lupus erythematosus (SLE) who are currently receiving cyclophosphamide. This study will also determine if RG2077 is effective in decreasing disease activity in these patients.

Study hypothesis: CTLA4-Ig mediates a T cell costimulatory blockade that effectively induces an antigen-specific nonresponsiveness in T cells.

DETAILED DESCRIPTION:
SLE is a chronic, inflammatory autoimmune disorder that may affect many organ systems, including the skin, joints, and internal organs. RG2077 has been studied for use in multiple sclerosis, another autoimmune disorder. This study will evaluate the safety and efficacy of RG2077 in SLE patients who are currently receiving cyclophosphamide.

This trial is composed of two parts. The first part is a dose-escalation study in which participants will receive one of two doses of RG2077 (0.2 mg/kg or 2 mg/kg); this part of the study will last 60 days. At screening, patients will have an IV catheter inserted into their arms for administration of cyclophosphamide and RG2077. Patients will also have medical and medication history assessments, a comprehensive physical exam, and blood and urine tests. There are 5 study visits for the first part of the trial; these will occur at screening, at study entry, and Days 1, 14, and 28. Selected visits will include physical exam, vital signs measurement, blood and urine tests, and disease activity assessment. At Days 7 and 60, patients will be contacted by phone to report their medication history and any adverse effects they have experienced.

The second part of the study will evaluate a single 10 mg/kg dose of RG2077; this part of the study will last 90 days. In the study, participants will be randomly assigned to one of two groups. At the start of the study, Group 1 participants will receive RG2077 and cyclophosphamide and Group 2 participants will receive cyclophosphamide only. There will be 9 study visits; these will occur at study screening, study entry, and Days 1, 4, 7, 14, 28, and 60. At selected visits, patients will undergo physical exam, vital signs measurement, blood tests and urine tests, and disease activity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE by American College of Rheumatology (ACR) criteria
* Concurrent treatment with intravenous cyclophosphamide (500 to 1000 mg/m2) for at least one of the following manifestations of lupus: World Health Organization (WHO) class III, IV, or V lupus nephritis; British Isles Lupus Assessment Group (BILAG) score of A for vasculitis; BILAG score of A for cytopenia; BILAG score of A for nervous system
* Stable medication regimen for at least 4 weeks prior to study entry
* Weight between 40 kg (88.2 lbs) and 125 kg (275.6 lb)
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Moderately severe anemia (hemoglobin less than 8 mg/dL)
* Neutropenia (absolute neutrophil count less than 1,500/mm3)
* Thrombocytopenia (platelets less than 50,000/mm3)
* Positive tuberculin (PPD) test without evidence of prior treatment or administration of bacille Calmette-Guérin (BCG) vaccine
* Active infections, including HIV and hepatitis B or C
* Receipt of a live vaccine within 3 months of study entry
* End-stage renal disease with creatinine clearance less than 20 ml/min/1.73 m2
* History of cancer. Patients with a history of carcinoma in situ and treated basal and squamous cell carcinomas are not excluded.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by the occurrence of adverse events | Throughout study

SECONDARY OUTCOMES:
Renal function | Throughout study
Lupus serology | Throughout study
SLE disease activity | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David Wofsy, MD, Study Chair — University of California, San Francisco; Betty Diamond, MD, Study Chair — Columbia University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Result] Davidson A, Diamond B, Wofsy D, Daikh D. Block and tackle: CTLA4Ig takes on lupus. Lupus. 2005;14(3):197-203. doi: 10.1191/0961203305lu2136oa. PMID 15807196
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- See also: Immune Tolerance Network (ITN) TrialShare: open public access to participant-level data available for this trial — http://www.itntrialshare.org
- Available data/document: Individual Participant Data Set: SDY798 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY798 — ImmPort study identifier is SDY798.
- Available data/document: Study protocol synopsis; -Study summary; -design; -adverse event; -Assessment; -Medications, -demographics; -study files: SDY798 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY798 — ImmPort study identifier is SDY798.
- Available data/document: Individual Participant Data Set: ITN002AI — http://www.itntrialshare.org/project/Studies/ITN002AIPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.
- Available data/document: Informed Consent Form: ITN002AI — http://www.itntrialshare.org/project/Studies/ITN002AIPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.
- Available data/document: Study synopsis, -schedule of events, -adverse events, et al.: ITN002AI — http://www.itntrialshare.org/project/Studies/ITN002AIPUBLIC/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.